CLINICAL TRIAL: NCT03407534
Title: Early Detection of Exocrine Pancreatic Insufficiency in Patients Presenting With Diarrhea and Bloating
Brief Title: Detection of Exocrine Pancreatic Insufficiency in Patients With Diarrhea and Bloating
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, M.D. Director of Advanced Endoscopy Assistant Professor of Medicine - Gastroenterology Section, Baylor College of Medicine
Other Study IDs: H-37932
Record Dates: First submitted 2017-07-28; First posted 2018-01-23 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Diarrhea; Exocrine Pancreatic Insufficiency; Abdominal Pain
Keywords: Exocrine; Pancreatic Insufficiency; Diarrhea; Bloating; Loose Stool
MeSH Terms: conditions — Diarrhea; Exocrine Pancreatic Insufficiency; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The prevalence of exocrine pancreatic insufficiency (EPI) among patients presenting with diarrhea and bloating as their chief complaints is not well studied. Diarrhea and or bloating can be due to different etiologies such as celiac disease and irritable bowel syndrome. However, concomitant EPI can exacerbate these conditions, or be the main cause of the symptoms. Furthermore, some of these diagnoses can be epiphenomena or consequences of EPI. The Investigators hypothesize that EPI will be detected in significant proportion of patients with bloating or diarrhea and that early detection and management of EPI can prevent unnecessary work up for other causes of diarrhea.

DETAILED DESCRIPTION:
Exocrine pancreatic insufficiency (EPI) diagnosis can be challenging due to several reasons. First, the main symptoms of EPI such as diarrhea, loose stool, bloating or weight loss have low specificity because they could be associated with many other conditions such as IBS or celiac disease. Second, EPI could be found concomitantly as an exacerbating factor with other causes of diarrhea and bloating leading to incomplete treatment and increased patient dissatisfaction due to partial resolution of symptoms. Although the prevalence of EPI in general population is not well known, a recent population study in 914 patients from Norway showed up to 10% prevalence of EPI using the measurement of fecal elastase-1 level in elderly. In another study, the prevalence of EPI diagnosed by low fecal elastase-1 in 314 patients with chronic diarrhea who satisfied the Rome II criteria for irritable bowel syndrome diarrhea (IBS-D) was 6.1%.Furthermore, an EPI prevalence of 4.4% (diagnosed by low fecal elastase-1) was documented in 90 patients who had serological and histological evidence of celiac disease. Interestingly, MRI was normal in all patients diagnosed with EPI in this study.

The gold standard tests for diagnosing EPI is three-day fecal fat quantification and determination of the coefficient of fat absorption. The patient is required to keep an intake of 100g of fat for five days and then collect feces for a time period of three days. Direct measurement of pancreatic function test with secreting stimulation is another sensitive test. . However these tests are cumbersome to apply to large number of patients with common complaints. Spot fecal elastase-1 measurement using enzyme linked immunosorbent assay (ELISA) has been shown to be highly sensitive and specific in diagnosing moderate to severe chronic pancreatitis in several studies. The favorable operating characteristics combined with the ease of using of the test makes it a good initial screening test for EPI.

Our preliminary data indicate that a large proportion (10 %) of patients with undiagnosed bloating and or diarrhea have EPI initially detected by low fecal elastase-1 and subsequently confirmed with Endoscopic Ultrasound and or direct measurement of pancreatic function tests. Therefore, Investigators propose to test the hypothesis that including fecal elastase-1 as part of the initial work-up for patients presenting with diarrhea and or bloating will identify patients who are confirmed EPI and may benefit from pancreatic enzyme replacement therapy and limit further unnecessary work up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old who presents to the gastroenterology clinic with main complaints of diarrhea
2. Patients aged 18-80 years old who presents to the gastroenterology clinic with main complaints of flatulence, and/or bloating
3. Patients with known IBS, microscopic colitis or celiac disease diagnosis will be included.
4. Patients on Diphenxoylate, loperamide or cholestyramin will be included.

Exclusion Criteria:

1. Known chronic pancreatitis, recurrent acute pancreatitis or autoimmune pancreatitis.
2. Known Pancreatic cancer
3. Prior History of distal pancreatictomy or Whipple surgery.
4. Prior history of gastric bypass surgery or any Roux en Y gastrojeujunal anastomosis.
5. Pregnant Patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population ages 18-80 will be recruited from St. Luke Baylor's Clinic during their clinic visit. Patients will receive full complete details about the research protocol and then will receive a consent form with all steps taken in details for the research. Participating in this research will be voluntary and if the patient decides to participate in the research they will need to sign and date the consent form. Patients to be recruited during the clinic visits are patients of the PI and/or of the Co-Investigators in this study.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2015-11; Primary Completion 2021-11-09 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Prevelance of Pancreatic Insufficency among patients that complain of symptoms of diarrhea and bloating | 4-6 Weeks
  1- Estimate the prevalence of the spectrum of EPI among patients presenting with diarrhea and bloating as chief complaints using fecal elastase-1 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Othman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Keihanian T, Agarwal S, Mansour N, Mercado M, El-Serag HB, Othman MO. Prevalence of Exocrine Pancreatic Insufficiency in Patients with Chronic Diarrhea. Saudi J Med Med Sci. 2025 Apr-Jun;13(2):99-105. doi: 10.4103/sjmms.sjmms_4_25. Epub 2025 Apr 21. PMID 40352337